CLINICAL TRIAL: NCT05173064
Title: Development and Randomized Controlled Trial of an AI-powered Technological Surrogate Physiotherapist (TSP) Dedicated to Quality Enhancement and Cost Reduction in Knee Osteoarthritis Exercise Rehabilitation
Brief Title: Effects of a Machine Learning-based Lower Limb Exercise Training System for Knee Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Feedback System
Record Dates: First submitted 2021-12-09; First posted 2021-12-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Pain; Knee Osteoarthritis
Keywords: knee pain, physical therapy, exercise
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The AI-powered Technological Surrogate Physiotherapist (Experimental): Participants will be required to perform three 30-minute exercise sessions per week for 12 weeks, with six exercises at any one time. During the exercise sessions, participants will receiveTechnological Surrogate Physiotherapist (TSP) support which will in particular leverage AI to offer innovative features and modules dedicated to enhancing exercise monitoring and supervision, real-time performance feedback, and self-assessment.
  Interventions: Device: The AI-powered Technological Surrogate Physiotherapist
- Face-to-face physiotherapist-supervised exercise program (Active Comparator): Participants will be required to visit a physiotherapist for usual face-to-face exercise therapy. Also, they will be required to perform three 30-minute home exercise sessions per week for 12 weeks. However, TSP will not be involved in this group.
  Interventions: Behavioral: Face-to-face physiotherapist-supervised exercise program
- The AI-powered Technological Surrogate Physiotherapist Plus Face-to-face physiotherapist-supervised (Experimental): Participants will receive an integrated intervention combining conventional physiotherapist-supervised sessions and TSP-supported home exercises (three 30-minute exercise sessions per week for 12 weeks).
  Interventions: Combination Product: The AI-powered Technological Surrogate Physiotherapist Plus Face-to-face physiotherapist-supervised exercise program

INTERVENTIONS:
Device: The AI-powered Technological Surrogate Physiotherapist — The AI-powered Technological Surrogate Physiotherapist will have three key features:
  1. Evidence-based exercise videos instructed by physical therapists
  2. Real-time movement feedback and performance score
  3. Exercise records.
  Arms: The AI-powered Technological Surrogate Physiotherapist
Behavioral: Face-to-face physiotherapist-supervised exercise program — Physiotherapists will give usual face-to-face therapy. The assessment of participants' exercise movements will only be achieved in the traditional manner during face-to-face exercise sessions - by physiotherapists' visual inspection of and professional judgement on postural alignment and effectiveness, with verbal instructions for posture correction. The features of real-time movement feedback and tracking of exercise progress will not be provided.
  Arms: Face-to-face physiotherapist-supervised exercise program
Combination Product: The AI-powered Technological Surrogate Physiotherapist Plus Face-to-face physiotherapist-supervised exercise program — This group will attend in-person group therapy sessions, while additionally completing weekly home exercise sessions using the TSP system.
  Arms: The AI-powered Technological Surrogate Physiotherapist Plus Face-to-face physiotherapist-supervised

SUMMARY:
The goal of the study is to confirm the idea of AI-powered Technological Surrogate Physiotherapist (TSP), by demonstrating its effectiveness and value as a new technology-based contribution to OA healthcare. Participants will be randomized to one of three groups: (1) the conventional PT group receiving the exercise program delivered through in-person sessions; (2) the AI-guided group following the program through the TSP after an initial PT session; or (3) the combined group receiving both in-person PT sessions and AI-guided home exercise. All individuals will take part in the study for 12 weeks, and data will be collected at baseline and 12 weeks after randomization.

DETAILED DESCRIPTION:
Knee pain, often caused by osteoarthritis, is a prevalent musculoskeletal disorder among older adults and significantly reduces physical function and quality of life. Exercise therapy has been shown to be an effective form of treatment for knee pain. However, the traditional delivery of exercise therapy requires that individuals attend clinics to participate in face-to-face exercise sessions, which can be expensive and inconvenient. In recent years, information technologies have been used to support the delivery of exercise programs. The programs have also shown great benefits in improving the management of knee pain. However, it remains a concern that physical therapists are not able to provide the patients with direct and immediate supervision when exercises are taken place remotely at home or in community centers, which can be detrimental to exercise performance and the management of knee pain.

Thus, the research team has developed a machine learning-based exercise training system to provide evidence-based lower limb exercise videos, real-time movement feedback, and tracking of exercise progress for older adults with knee pain. In this study, a 12-week randomized controlled non-inferiority trial will be conducted to examine the effects of AI-powered Technological Surrogate Physiotherapist, comparing with the effects of the group receiving in-person sessions and effects of the combined group receiving both.

ELIGIBILITY:
Inclusion Criteria:

Participants will be recruited if they

* age ≥ 50 years,
* report having pain in or around the knee for more than 12 weeks and on most days of the previous month,
* report being diagnosed with knee OA by a physician, have physician-diagnosed knee OA in the medical record, or have radiographic evidence of grade 2 to 3 knee OA on the Kellgren-Lawrence scale in the posteroanterior and/or skyline view or the presence of lateral/posterior osteophytes (the X-rays will be read and classified by our orthopaedic surgeons collaborators to decide on each patient's eligibility to be included in the study),
* are willing and physically and cognitively able to perform (technology-supported) exercises required in the study protocol
* have normal or corrected to normal vision,
* are able to speak and read Chinese,
* are able to provide written informed consent.

Exclusion Criteria:

Individuals will be excluded if they have

* history of knee or hip replacement surgery,
* non-ambulatory status,
* systemic inflammatory arthritis (e.g., gout),
* history of trauma (e.g., fractures around the knee, dislocation, and sprains or tears of soft tissues, like ligaments) or surgical arthroscopy of either knee within the past 6 months,
* intra-articular injection to the knee within the past 6 months,
* cognitive impairment,
* involvement in a similar study in the past 6 months,
* recent or imminent surgery (within 12 weeks),
* medical co-morbidities that preclude participation in exercise.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in knee pain as assessed by a 11-point numerical pain rating scale as recommended by the OARSI | From baseline to 12 weeks
  0 represents no pain and 10 represents the worst possible pain.
Changes in physical function as assessed by the Knee Injury and Osteoarthritis Outcome Score (KOOS) physical function sub-scale | From baseline to 12 weeks
  The scale regards the degree of difficulty in performing usual daily activities and higher level activities that involve physical function of the knee. Each item will be rated on a 5-point Likert scale ranging from 'None' (i.e., no difficulty) to 'Extreme' (i.e., extreme difficulty), based on which a normalized total score will be calculated (0 indicating extreme symptoms and 100 indicating no symptoms).

SECONDARY OUTCOMES:
Changes in physical function as assessed by 30-second chair-stand test | From baseline to 12 weeks
  30-second chair stand test (30CST), which measures the number of stands the participant can complete in 30 sec, will be used to assess the general leg strength and functional performance.
Changes in physical function as assessed by timed up-and-go test | From baseline to 12 weeks
  Timed up and go (TUG) test, which measures the time it takes the participant to standup from the chair, walk 3 meters, walk back to the chair, and sit down, will be used to assess functional mobility.
Changes in physical function as assessed by maximal isometric strength of the quadriceps and hamstrings | From baseline to 12 weeks
  The participant will be instructed to maximally extend/flex each knee for 3 trials, 3 sec each, with a 1-minute rest in between. Verbal encouragement will be given in each trial to ensure the participant makes the maximum effort. The highest force of each muscle in the three trials will be used for data analysis.
  After each test trial, the severity of pain experienced by the participant during the trial will be assessed using the 11-point numerical pain rating scale.
Changes in physical function as assessed by active and passive ranges of motion of the hip and knee joints | From baseline to 12 weeks
  Active and passive ranges of motion of the hip and knee joints will be assessed using a goniometer.
Changes in health-related quality of life assessed by the Chinese version of the 36-item Short Form Survey (SF-36) | From baseline to 12 weeks
  Health-related quality of life will be assessed using the Chinese version of the 36-item Short Form Survey (SF-36).
Exercise adherence | From baseline to 12 weeks
  Exercise adherence will be indicated by the proportion of sessions and proportion of exercises performed which will be recorded by the TSP system (only for intervention group) and by participants and researchers using a log book.
Satisfaction with the therapeutic exercise training | From baseline to 12 weeks
  It will be rated by participants using a 7-point Likert scale with anchors of 'Extremely unsatisfied' and 'Extremely satisfied'.
Convenience in terms of location and time for accessing the exercise therapy | From baseline to 12 weeks
  It will be assessed on an 11-point numerical rating scale, with 0 representing 'Extremely inconvenient' and 10 representing 'Extremely convenient'.

CONTACTS AND LOCATIONS:
Locations (1):
- 826, Haking Wong Building, Pokfulam, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts JM, Wilson K. Effect of stretching duration on active and passive range of motion in the lower extremity. Br J Sports Med. 1999 Aug;33(4):259-63. doi: 10.1136/bjsm.33.4.259. PMID 10450481
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Hinman RS, Kimp AJ, Campbell PK, Russell T, Foster NE, Kasza J, Harris A, Bennell KL. Technology versus tradition: a non-inferiority trial comparing video to face-to-face consultations with a physiotherapist for people with knee osteoarthritis. Protocol for the PEAK randomised controlled trial. BMC Musculoskelet Disord. 2020 Aug 7;21(1):522. doi: 10.1186/s12891-020-03523-8. PMID 32767989
- [Background] Lam CL, Tse EY, Gandek B, Fong DY. The SF-36 summary scales were valid, reliable, and equivalent in a Chinese population. J Clin Epidemiol. 2005 Aug;58(8):815-22. doi: 10.1016/j.jclinepi.2004.12.008. PMID 16018917
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] McAlindon TE, Driban JB, Henrotin Y, Hunter DJ, Jiang GL, Skou ST, Wang S, Schnitzer T. OARSI Clinical Trials Recommendations: Design, conduct, and reporting of clinical trials for knee osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):747-60. doi: 10.1016/j.joca.2015.03.005. PMID 25952346
- [Background] McAlindon TE, Cooper C, Kirwan JR, Dieppe PA. Knee pain and disability in the community. Br J Rheumatol. 1992 Mar;31(3):189-92. doi: 10.1093/rheumatology/31.3.189. PMID 1540789
- [Background] Cottrell E, Roddy E, Foster NE. The attitudes, beliefs and behaviours of GPs regarding exercise for chronic knee pain: a systematic review. BMC Fam Pract. 2010 Jan 18;11:4. doi: 10.1186/1471-2296-11-4. PMID 20082694
- [Background] Hurley MV, Walsh NE, Mitchell HL, Pimm TJ, Patel A, Williamson E, Jones RH, Dieppe PA, Reeves BC. Clinical effectiveness of a rehabilitation program integrating exercise, self-management, and active coping strategies for chronic knee pain: a cluster randomized trial. Arthritis Rheum. 2007 Oct 15;57(7):1211-9. doi: 10.1002/art.22995. PMID 17907147
- [Background] Hurley MV, Walsh NE, Mitchell H, Nicholas J, Patel A. Long-term outcomes and costs of an integrated rehabilitation program for chronic knee pain: a pragmatic, cluster randomized, controlled trial. Arthritis Care Res (Hoboken). 2012 Feb;64(2):238-47. doi: 10.1002/acr.20642. PMID 21954131
- [Background] Chen T, Or CK, Chen J. Effects of technology-supported exercise programs on the knee pain, physical function, and quality of life of individuals with knee osteoarthritis and/or chronic knee pain: A systematic review and meta-analysis of randomized controlled trials. J Am Med Inform Assoc. 2021 Feb 15;28(2):414-423. doi: 10.1093/jamia/ocaa282. PMID 33236109
- [Background] Hay EM, Foster NE, Thomas E, Peat G, Phelan M, Yates HE, Blenkinsopp A, Sim J. Effectiveness of community physiotherapy and enhanced pharmacy review for knee pain in people aged over 55 presenting to primary care: pragmatic randomised trial. BMJ. 2006 Nov 11;333(7576):995. doi: 10.1136/bmj.38977.590752.0B. Epub 2006 Oct 20. PMID 17056608